CLINICAL TRIAL: NCT06263764
Title: The Effect of Listening to Qur'an Recital on Quality of Life in Systemic Lupus Erythematosus Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dr. dr. Alvina Widhani, Sp.PD, KAI, Staff of Allergy Immunology Division, Department of Internal Medicine, Faculty of Medicine Universitas Indonesia, Indonesia University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 23-11-1954
Record Dates: First submitted 2024-02-08; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Quality of Life
Keywords: Quran Recital; Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qur'an Arm (Experimental): Participants in the intervention group will be asked to listen to a Qur'an recital by Surah Ar-Rahman using an MP3 player twice a day for a minimum of 15 minutes each for 40 days.
  The participants will listen to the same Qur'an recital (recited by Freed Ghalib) using the same MP3 player.
  Interventions: Other: Listening to Qur'an Recital
- Control Arm (No Intervention): The control group will not receive any specific intervention and will continue with their usual routine

INTERVENTIONS:
Other: Listening to Qur'an Recital — Listening to Surah Ar Rahman twice a day for minimum 15 minutes each for 40 days
  Arms: Qur'an Arm

SUMMARY:
The goal of this quasi-experimental study is to evaluate the effect of listening to the Qur'an recital on quality of life among systemic lupus erythematosus patients. There will be intervention and control groups. Before the intervention, the quality of life of participants will be assessed using the Lupus-QoL questionnaire. After the baseline assessment, participants in the intervention group will be asked to listen to a Qur'an recital by Surah Ar-Rahman using an MP3 player twice a day for a minimum of 15 minutes each for 40 days. The control group will not receive any specific intervention and will continue with their usual routine. After the 40-day intervention period, the quality of life of participants in both groups will be assessed using the Lupus-QoL questionnaire. The results will be analyzed to determine if there is a significant improvement in quality of life. Besides, potential confounding factors such as SLE clinical manifestations, disease activity, pharmacologic treatment regimen, anxiety/depression, comorbidities, age, and economic status will also be collected before and after intervention to evaluate its effect on the quality of life.

DETAILED DESCRIPTION:
Subjects who meet the eligibility criteria will be classified into intervention and control groups based on their Qur'an listening routine. Those who listen to the Qur'an less than once a week will be included in the control group. On the other hand, those who listen to the Qur'an once or more a week will be included in the intervention group. Before the intervention, we will also evaluate the potential confounding factors in each respondent that could affect quality of life, such as SLE clinical manifestations, disease activity, pharmacologic treatment regimen, anxiety or depression, comorbidities, and economic status.

Subjects in the intervention group will be asked to listen to the Al Qur'an recital (QS. Ar-Rahman) with a minimum duration of 15 minutes each, twice every day for 40 days, through an MP3 player using a headset or earphone. They will listen to the same Qur'an recital that is recited by Freed Ghalib. To ensure the respondents listen to the Qur'an recital Surah Ar-Rahman, the researcher will call and message via the Whats App application to research subjects every day for reminding. Respondents are also given a checklist card that will be filled out each time they are finished listening to the Qur'an recital. The control group will be asked not to change their habits of listening to or reading the Qur'an during this period. In addition, both the intervention and control groups will also be asked to inform the researchers if they read the Qur'an during the intervention or monitoring period.

ELIGIBILITY:
Inclusion Criteria:

* Systemic Lupus Erythematosus Patients based on EULAR/ACR 2019 diagnostic criteria,
* Female aged ≥ 18 years old,
* Muslim (follower of the religion of Islam),
* Have no auditory problems,
* Received a steroid dose ≤ 20 mg/day equivalent to prednisone,

Exclusion Criteria:

* Cannot read or write,
* Using drugs that affect the work of the central nervous system,
* Not willing to take part in research.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 70 (Estimated)
Dates: Start 2024-02-12 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Difference in Quality of Life Pre and Post Intervention | 40 days
  Difference in quality of life score (Lupus-QoL score)

CONTACTS AND LOCATIONS:
Overall Officials: Rudi Putranto, PhD, Study Director — Department of Internal Medicine, Faculty of Medicine Universitas Indonesia; Sukamto Koesnoe, PhD, Study Director — Department of Internal Medicine, Faculty of Medicine Universitas Indonesia; Alvina Widhani, PhD, Principal Investigator — Department of Internal Medicine, Faculty of Medicine Universitas Indonesia; Karina Wijayanti, MD, Principal Investigator — Department of Internal Medicine, Faculty of Medicine Universitas Indonesia
Locations (1):
- Faculty of Medicine Universitas Indonesia -Cipto Mangunkusumo Hospital, Jakarta, Indonesia, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rafique R, Anjum A, Raheem SS. Efficacy of Surah Al-Rehman in Managing Depression in Muslim Women. J Relig Health. 2019 Apr;58(2):516-526. doi: 10.1007/s10943-017-0492-z. PMID 28900859